CLINICAL TRIAL: NCT02516163
Title: A Prospective, Non-randomized,Study of the Clinical Outcomes of Participants That Receive the Stryker Triathlon Total Knee System for Total Knee Arthroplasty Implanted Using ShapeMatch® Cutting Guides: Sub-Study A
Brief Title: Stryker Triathlon Total Knee System for Total Knee Arthroplasty Implanted Using Shapematch Cutting Guides:Sub-Study A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker South Pacific (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TriShapeMatch-10_Substudy A
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-09

CONDITIONS: Arthroplasties, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shapematch Cutting Guides (Other): The ShapeMatch® Cutting Guides are intended to be used as patient-specific surgical instrumentation to assist in the positioning of knee arthroplasty components intra-operatively and in guiding the marking of bone before cutting.
  They are intended for single use only.
  Interventions: Device: Shapematch Cutting Guides

INTERVENTIONS:
Device: Shapematch Cutting Guides — Participants will undergo pre-operative assessment using MRI of the affected limb. At the time of surgery, a repeated-measures methodology will be implemented in which the position of the femoral and tibial cutting guides will be measured using the Navigation system. The same surgeon will position each cutting guide a total of 3 times for each patient. Multiple participants will be assessed by each surgeon. No bone cuts will take place using the patient-specific cutting guides. After the study-specific measurements have been taken, the total knee procedure will resume using the Navigation system and associated instruments. No post-operative evaluations will be undertaken as part of this sub-study

SUMMARY:
This is a prospective, non-randomized, study of the clinical outcomes of participants that receive the Stryker Triathlon® Total Knee System for Total Knee Arthroplasty implanted using ShapeMatch® Cutting Guides.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, study of the clinical outcomes of participants that receive the Stryker Triathlon® Total Knee System for Total Knee Arthroplasty implanted using ShapeMatch® Cutting Guides. Sub-study A aims to quantify the reproducibility of intra-operatively positioning the cutting guides onto the affected femoral and tibial joint surfaces.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or non-pregnant female between the ages of 50-90.
* The patient requires a primary total knee replacement and is indicated for computer-assisted surgery.
* The patient has a primary diagnosis of osteoarthritis (OA).
* The patient has intact collateral ligaments.
* The patient is able to undergo MRI scanning of the affected limb.
* The patient has signed the study specific, HREC-approved, Informed Consent document.
* The patient is willing and able to comply with the specified pre-operative and post-operative clinical and radiographic evaluations.

Exclusion Criteria:

* The patient has a history of total, unicompartmental reconstruction or fusion of the affected joint.
* The patient has had a high tibial osteotomy or femoral osteotomy.
* The patient is morbidly obese (BMI ≥ 40).
* The patient has a deformity which will require the use of stems, wedges or augments in conjunction with the Triathlon Total Knee System.
* The patient has a varus/valgus malalignment ≥ 15° (relative to mechanical axis).
* The patient has a fixed flexion deformity ≥ 15°.
* The patient has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* The patient has a systemic or metabolic disorder leading to progressive bone deterioration.
* The patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements.
* The patient has a cognitive impairment, an intellectual disability or a mental illness.
* The patient is pregnant.
* The patient has metal hardware present in the region of the hip, knee or ankle (as this is known to create geometrical distortion in the region of the implant).
* The patient has any known contraindications for undergoing assessment by MRI (e.g. ferrous implants, metallic clips, magnetically activated implanted devices such as cardiac pacemakers, etc).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 55 knees enrolled - 3 censored from analysis due to major protocol deviations = 52 knees in study analysis.
Groups:
- Shapematch Cutting Guides: The ShapeMatch® Cutting Guides are patient-specific surgical instruments to assist in the positioning of knee arthroplasty components intra-operatively and in guiding the marking of bone before cutting.They are single use only. Participants undergo pre-operative assessment using MRI of the affected limb. At the time of surgery, a repeated-measures methodology is implemented in which the position of the femoral and tibial cutting guides is measured using the Navigation system. The same surgeon will position each cutting guide a total of 3 times for each patient. No bone cuts will take place using the patient-specific cutting guides. After the study-specific measurements have been taken, the total knee procedure will resume using the Navigation system and instruments. No post-operative evaluations will be undertaken as part of this sub-study.
Period: Overall Study
Arm/Group | Shapematch Cutting Guides
Started | 52
Completed | 24
Not Completed | 28
Not completed — Withdrawal by Subject | 1
Not completed — Failed MRI/incorrect MRI protocol | 11
Not completed — Unfit/delay in surgery | 3
Not completed — Use of incorrect measurement technique | 5
Not completed — Data not recorded | 2
Not completed — MRI contraindication exclusion | 6

BASELINE CHARACTERISTICS:
Population: Baseline measurements are available only for the 24 participants who completed the study.
Arm/Group | Shapematch Cutting Guides
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Region of Enrollment [Number; unit: participants]
  Australia | 24

OUTCOME MEASURES:

1. Primary Outcome: Repeatability of Cutting Guide Position
Description: Repeatability of cutting guide position on the distal femur and proximal tibia assessed by repeated measures using computer navigation system for total knee replacement, assessed intra-operatively. Placement of the cutting guides by the surgeon was determined by recording the position of the cutting guide when placed by the same surgeon multiple times. The intraclass correlation coefficient (ICC) was calculated for each positioning parameter. This included femoral and tibial varus/valgus,flexion/extension, medial resection, lateral resection and rotation. ICC agreement categories:>0.75 excellent agreement; 0.75-0.4 good or fair agreement; <0.4 poor agreement.
Time Frame: Intraoperative - participants were followed for the duration of the operation, an average of 1 hour and 50 minutes.
Measure: Number (95% Confidence Interval); unit: intraclass correlation coefficient (ICC)
Units Other Than Participants: Knees
Arm/Group | Shapematch Cutting Guides
Number analyzed (Participants) | 24
Number analyzed (Knees) | 24
intraclass correlation coefficient (ICC)
  Femur varus/valgus ICC | 0.990 [0.980 to 0.995]
  Femur flexion/extension ICC | 0.963 [0.929 to 0.983]
  Femur medial resection ICC | 0.936 [0.879 to 0.970]
  Femur lateral resection ICC | 0.910 [0.832 to 0.957]
  Femur rotation ICC | 0.993 [0.987 to 0.997]
  Tibia varus/valgus ICC | 0.994 [0.989 to 0.997]
  Tibia flexion/extension ICC | 0.961 [0.925 to 0.982]
  Tibia medial resection ICC | 0.889 [0.795 to 0.946]
  Tibia lateral resection ICC | 0.940 [0.887 to 0.972]
  Tibia rotation ICC | 0.997 [0.995 to 0.999]

ADVERSE EVENTS:
Time Frame: Intraoperative- participants were followed for the duration of the operation, an average of 1 hour and 50 minutes.
Description: Elective procedures not included.e.g.non-study joint replacement/revision, rotator cuff repair,carpal tunnel release,cataract,intra-ocular & bunion procedures,total shoulder repair,laminectomy,microdiscectomy,breast reduction,cervical spine fusion,& mid/flat-foot surgery.Industry standard AE terms not used;specific AE terms not used for all AEs.
Groups:
- Shapematch Cutting Guides: The ShapeMatch® Cutting Guides are intended to be used as patient-specific surgical instrumentation to assist in the positioning of knee arthroplasty components intra-operatively and in guiding the marking of bone before cutting.
  They are intended for single use only.
  Shapematch Cutting Guides: Participants will undergo pre-operative assessment using MRI of the affected limb. At the time of surgery, a repeated-measures methodology will be implemented in which the position of the femoral and tibial cutting guides will be measured using the Navigation system. The same surgeon will position each cutting guide a total of 3 times for each patient. Multiple participants will be assessed by each surgeon. No bone cuts will take place using the patient-specific cutting guides. After the study-specific measurements have been taken, the total knee procedure will resume using the Navigation system instruments. No post-operative evaluations will be undertaken as part of this sub-study
Arm/Group | Shapematch Cutting Guides
Serious Adverse Events (participants affected / at risk) | 2/52
Other Adverse Events (participants affected / at risk) | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shapematch Cutting Guides (N=52)
non-operative site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Operative site (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Discloser must give at least 40 days notice to Sponsor including a copy of the proposed publication. The Sponsor can then provide comments (which Discloser is not bound to follow), request delay of publication by no more than 120 days to allow for Sponsor to protect its intellectual property, or request that the Discloser remove certain proprietary or confidential information from the study (other than the results of the study).